CLINICAL TRIAL: NCT06173375
Title: Comparative Effectiveness Pilot Trial of Mailed Cologuard Outreach to Mailed FIT Outreach
Brief Title: Head to Head Pilot Trial of Mailed Cologuard to Mailed FIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Joshua Demb, PhD, MPH, Postdoctoral Scholar, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 803124
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer
Keywords: screening; early detection; stool blood test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Two-arm intervention trial comparing mailed Cologuard outreach (intervention) to mailed FIT outreach (control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mailed Cologuard Outreach (Experimental): Receipt of mailed Cologuard test for colorectal cancer screening to be completed and returned by participant. If test is negative, participant will be advised to undergo another test in 3 years. If test is positive, participant will be advised to schedule colonoscopy for further testing.
  Interventions: Diagnostic Test: Cologuard
- Mailed Fecal immunochemical test Outreach (Active Comparator): Receipt of mailed FIT for colorectal cancer screening to be completed and returned by participant. If test is negative, participant will be advised to undergo another test in 1 year. If test is positive, participant will be advised to schedule colonoscopy for further testing.
  Interventions: Diagnostic Test: Fecal Immunochemical Test

INTERVENTIONS:
Diagnostic Test: Cologuard — Multi-target stool DNA test for colorectal cancer screening implemented by Exact Sciences. Cologuard has 94% sensitivity and 87% specificity to detect colorectal cancer.
  Arms: Mailed Cologuard Outreach
Diagnostic Test: Fecal Immunochemical Test — Stool blood test for colorectal cancer screening. FIT has 75% sensitivity and 90% specificity to detect colorectal cancer.
  Other Names: OC-Sensor Test
  Arms: Mailed Fecal immunochemical test Outreach

SUMMARY:
The objective of this pilot study is to compare the effectiveness of mailed outreach of two stool based tests, Cologuard and the fecal immunochemical test (FIT) in screening eligible adults ages 45-49 receiving care at the University of California San Diego Health system.

DETAILED DESCRIPTION:
Adults ages 45-49 who are insured, deemed average risk and not currently up to date with colorectal cancer screening will be enrolled. Eligible participants will be randomized to either mailed Cologuard outreach, facilitated by Exact Sciences or mailed FIT outreach. Colorectal cancer screening completion within 3 months will be measured as the primary outcome, in addition to secondary recruitment and intervention-based feasibility outcomes to demonstrate the potential for a larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 45-49 with EHR documentation indicating that the patient has an assigned primary care provider at UCSD Health
* ≥1 UCSD Health System health visit within the last year
* Resides in San Diego or Imperial County
* Currently not up to date with CRC screening
* Insured by private, public or other health insurance.

Exclusion Criteria:

* Up-to-date with screening
* Prior history of colonic disease, including inflammatory bowel disease, one or more colorectal neoplastic polyps (i.e., adenomas) or colorectal cancer.
* Prior history of colectomy
* Lack of health insurance

Ages: 45 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Colorectal cancer screening completion | Within 3 months of randomization
  The proportion of individuals who complete any colorectal cancer screening test recommended by US Preventive Services Task Force (colonoscopy, FIT, Cologuard, Sigmoidoscopy or CT Colonography)
Proportion of Abnormal stool blood test results | Within 3 months of randomization
  Among those completing designed interventions (Cologuard or FIT), the proportion of test results yielding an abnormal result.
Proportion of Follow-up colonoscopy after abnormal stool blood test result | Within 6 months after stool blood test completion
  Among those with positive stool blood test results, the proportion who complete diagnostic follow-up colonoscopy

SECONDARY OUTCOMES:
Number of participants opting out of the pilot | Within 3 months of randomization
  Measurement of feasibility of pilot
Number of participants with undeliverable FIT or Cologuard tests (mail fail rate) | Within 3 months of randomization
  Measurement of feasibility of mailed outreach
Number of Adenomas detected | Within 6 months after screening test completion
  Measurement of number of adenomas detected during study period
Number of sessile serrated lesions detected | Within 6 months after screening test completion
  Measurement of number of sessile serrated lesions detected during study period
Number of colorectal cancer cases detected | Within 6 months after screening test completion
  Number of colorectal cancers detected during study period

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Demb, PhD, Principal Investigator — Postdoctoral Researcher
Locations (1):
- University of California San Diego, La Jolla, California, United States